CLINICAL TRIAL: NCT07280637
Title: Treatment of Periocular Wrinkles With the Active Ingredients PDRN, Hyaluronic Acid and Niacinamide, Applied by Needling or Microneedling: Randomized Clinical Trial"
Brief Title: Regenarative Treatment of Periocular Wrinkles With PDRN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Taubate (Other)
Collaborators: Cavalca & Cortelli private research center (Unknown)
Responsible Party: Principal Investigator, Jose Roberto Cortelli, Titular Professor, University of Taubate
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE77259324.6.0000.5501
Record Dates: First submitted 2025-11-27; First posted 2025-12-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Skin Wrinklings
MeSH Terms: interventions — Injections, Intradermal

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, parallel groups
Who Masked: Outcomes Assessor
Masking Description: statistics
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradermotherapy (Experimental): polydeoxyribonucleotides (PDRN) 0.5% PDRN combined with 2% hyaluronic acid and 0.1% niacinamide delivered by intradermal injection
  Interventions: Procedure: Intradermal injection
- Microneedling (Active Comparator): polydeoxyribonucleotides (PDRN) 0.5% PDRN combined with 2% hyaluronic acid and 0.1% niacinamide delivered by micro needling
  Interventions: Procedure: Micro needling

INTERVENTIONS:
Procedure: Intradermal injection — three periorbital intradermal injection sessions, at 30-day intervals, of polydeoxyribonucleotides (PDRN) 0.5% combined with 2% hyaluronic acid and 0.1% niacinamide
  Other Names: Intradermotherapy
  Arms: Intradermotherapy
Procedure: Micro needling — three periorbital micro needling sessions, at 30-day intervals, with polydeoxyribonucleotides (PDRN) 0.5% combined with 2% hyaluronic acid and 0.1% niacinamide
  Arms: Microneedling

SUMMARY:
This randomized clinical trial aims to compare two application techniques-needling (intradermal needling) and microneedling-for the delivery of an active-ingredient formulation containing 0.2% polynucleotides (PDRN), 2% hyaluronic acid, and 0.1% niacinamide for the treatment of periocular wrinkles related to aging.

DETAILED DESCRIPTION:
Facial aging in the periocular region results from cumulative sun exposure, reduced dermal thickness, and repetitive muscular contraction, contributing to wrinkle formation and loss of skin quality. Polynucleotides (PDRN) have been reported as cellular-regeneration agents with potential to improve skin texture, hydration, and tissue recovery. The present study evaluates the clinical efficacy of a formulation composed of 0.2% PDRN, 2% hyaluronic acid, and 0.1% niacinamide, delivered by two minimally invasive techniques: needling (intradermal needling) and microneedling.

Twenty four participants will be randomly allocated (1:1) into two treatment arms: needling (n=12) or microneedling (n=12). Each participant will receive three treatment sessions spaced 30 days apart, with a total volume of 1 mL applied per session. Standardized 3D facial imaging (Vectra system) will be used to assess periocular wrinkle severity (0-100%), Glogau's photoaging scale (scores 1 - 4), epigenetic markers along with skin-quality parameters, pigmentation, and inflammatory response at baseline and at 30 and 180 days following the first session. Intra-group and inter-group comparisons will be conducted using a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Glogau II and III
* Fitzpatrick II and III

Exclusion Criteria:

* Pregnancy
* immune diseases
* tabagism
* aesthetics facial treatment in the past 6 months

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
severity of periocular wrinkles | baseline vs. 30 days
  changes in the severity (0-100%) of periocular wrinkles measured in 3-dimensional (3D) facial photographs

SECONDARY OUTCOMES:
Glogau's facial photoaging scale | Baseline vs. 6 months
  Changes in Glogau scores (ranging 1 - 4); higher scores indicate worse outcome
LINE-1 | baseline vs. 30 days
  Changes in DNA methylation (5-meC), hydroxymethylation (5-hmeC) and 5-meC/5-hmeC ratio in the promoter region of LINE-1 elements
LINE-1 | baseline vs. 6 months
  Changes in DNA methylation (5-meC), hydroxymethylation (5-hmeC) and 5-meC/5-hmeC ratio in the promoter region of LINE-1 elements
severity of periocular wrinkles | Baseline vs. 6 months
  changes in the severity (0-100%) of periocular wrinkles measured in 3-dimensional (3D) facial photographs

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Cortelli, doctorate, Principal Investigator — Univeristy of Taubate
Locations (1):
- Cavalca & Cortelli private research center, Taubaté, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Only group and codified data will be shared with study staff.